CLINICAL TRIAL: NCT03710941
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Intravenously Administered REGN2477+REGN1033 in Patients With Sporadic Inclusion Body Myositis
Brief Title: Safety and Efficacy of REGN2477+REGN1033 in Patients With Sporadic Inclusion Body Myositis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to an internal decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R2477-1033-sIBM-1828; 2018-002853-31 (EudraCT Number)
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Sporadic Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN2477+REGN1033 (Experimental): Single, sequential, repeat-dose IV or matching placebo
  Interventions: Drug: REGN2477+REGN1033
- Placebo (Experimental): Single, sequential, repeat-dose IV
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: REGN2477+REGN1033 — Single, sequential, repeat-dose Intravenous (IV) or matching placebo
  Arms: REGN2477+REGN1033
Drug: Matching placebo — Single, sequential, repeat-dose Intravenous (IV)
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of REGN2477+REGN1033 in combination on total lean mass, as measured by Dual-energy X-ray absorptiometry (DXA) in patients with sporadic inclusion body myositis (sIBM).

The secondary objectives of the study are:

* To evaluate the efficacy of REGN2477+REGN1033 on the IBM-Functional Rating Scale (IBM-FRS)
* To evaluate the efficacy of REGN2477+REGN1033 on the sIBM Physical Functioning Assessment (sIFA)
* To evaluate the safety and tolerability of REGN2477+REGN1033
* To evaluate the effects of REGN2477+REGN1033 on body composition by DXA, including appendicular lean mass and total fat mass
* To evaluate the efficacy of REGN2477+REGN1033 on measures of muscle performance and physical function
* To evaluate the efficacy of REGN2477+REGN1033 on patient reported outcome measures including the fear of falling, falls and near falls, and health-related quality of life
* To evaluate the pharmacokinetic(s) (PK) profile of REGN2477+REGN1033, including functional REGN2477 and functional REGN1033 concentrations in serum over time
* To evaluate the immunogenicity of REGN2477+REGN1033

ELIGIBILITY:
Key Inclusion Criteria:

* Men and postmenopausal* women
* Diagnosed with sIBM based on the European Neuromuscular Centre (ENMC) IBM Research Diagnostic Criteria
* Ability to walk ≥150 meters, with or without a walking aid such as cane or walker, in 6 minutes.
* Ability to climb 4 steps of stairs unassisted (may use handrails)
* Willing and able to comply with clinic visits and study-related procedures

Key Exclusion Criteria:

* Other neurological conditions (eg, hemiplegia post stroke, Parkinson's) or musculo-skeletal conditions (eg, severe osteoarthritis) causing mobility impairment
* Mini-Mental State Examination (MMSE) score <24
* Ongoing, chronic, high-dose (>20 mg prednisone equivalent per day), systemic corticosteroid therapy within 6 weeks prior to screening.
* Any condition that precludes adequate intake of energy and protein; malnutrition; presence of an eating disorder.
* Unintentional weight loss of ≥10% in the past 6 months (patient-reported)
* Hospitalization for heart failure in last year or New York Heart Association Class 4
* History of hypertrophic cardiomyopathy
* Any drugs known to influence muscle mass and performance such as anabolic steroids or growth hormone within 6 weeks prior to screening
* Unable to fit on the site's DXA scanner table, within borders for scanning of total lean mass

Note: Other protocol Inclusion/Exclusion criteria apply

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-19 (Estimated); Primary Completion 2020-08-27 (Estimated); Study Completion 2020-11-05 (Estimated)

PRIMARY OUTCOMES:
Percent change in total lean mass as measured by dual-energy X-ray absorptiometry (DXA) | Up to Week 20

SECONDARY OUTCOMES:
Change in the Inclusion Body Myositis-Functional Rating Scale (IBM-FRS) | Up to Week 26
Change in the Sporadic inclusion body myositis (sIBM) Physical Functioning Assessment (sIFA) | Up to Week 26
Incidence and severity of treatment-emergent adverse events (TEAEs) | Up to Week 30
Percent change in total and regional body composition (including lean mass and fat mass) as measured by DXA | Up to Week 30
Absolute change in total and regional body composition (including lean mass and fat mass) as measured by DXA | Up to Week 30
Change in the 1-repetition maximum (1-RM) chest press strength | Up to Week 26
Change in hand-grip strength as measured by dynamometry | Up to Week 26
Change in distance walked in the 6-minute walk test (6MWT) | Up to Week 26
Change in time to complete the 10-meter walk test (10MWT) | Up to Week 26
Change in instrumented stair climb power | Up to Week 26
Change in instrumented, sensor-based sit-to-stand test time | Up to Week 26
Change in fear of falling as measured via the Falls Efficacy Scale-International (FES-I) | Up to Week 30
Change in Patient Global Impression of Severity assessments (PGIS/PGIC) | Up to Week 30
Change in Patient Global Impression of Change Items assessments (PGIS/PGIC) | Up to Week 30
Change in Clinician Global Impression of Severity assessments (CGIS/CGIC) | Up to Week 30
Change in Clinician Global Impression of Change Items assessments (CGIS/CGIC) | Up to Week 30
Change in 36-item Short Form Health Survey (SF-36), including the Physical Function Items (PF-10) and the Vitality Scale of the SF-36 | Up to Week 30
Change in Thigh muscle volume as measured by MRI (sub-study) | Up to Week 30
Frequency of falls and near-falls as measured by the Hopkins Falls Grading Scale | Up to Week 30
Pharmacokinetics (PK) profile of REGN2477 | Up to Week 30
  Assessed via serum concentration of REGN2477 over time
Pharmacokinetics (PK) profile of REGN1033 | Up to Week 30
  Assessed via serum concentration of REGN1033 over time
Immunogenicity of REGN2477+REGN1033 | Up to Week 30
  As determined by the presence or absence of anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals